CLINICAL TRIAL: NCT02416830
Title: Worldwide Therapeutic Embolization Cohort Post Market Registry
Acronym: EmboReg
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: EmboCoH (Other)
Responsible Party: Sponsor
Other Study IDs: embocohort
Record Dates: First submitted 2015-03-31; First posted 2015-04-15 (Estimated); Last update posted 2015-04-15 (Estimated); Status verified 2015-04

CONDITIONS: Aortic; Peripheral; and Visceral Artery Aneurysms
Keywords: embolization; visceral Aneurysms; Prospective Registry

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this cohort post market registry is to collect data and create a global database on use of embolization devices and embolization procedures outcome. The data collected in the cohort will serve a scientific purpose to acquire better insight in embolization procedures. This will be achieved by publications in Scientific Journals and by presentations at scientific meetings. Additionally it will support the industry on creating a better overview of the products used to maintain and enhance the clinical efficacy of the used devices. The cohort post market registry represents a novel approach in a way of allowing Clinicians to generate reports based on an evolving controlled and well organized database

DETAILED DESCRIPTION:
INTRODUCTION

Purpose:

The purpose of this cohort post market registry is to collect data and create a global database on use of embolization devices and embolization procedures outcome. The data collected in the cohort will serve a scientific purpose to acquire better insight in embolization procedures. This will be achieved by publications in Scientific Journals and by presentations at scientific meetings. Additionally it will support the industry on creating a better overview of the products used to maintain and enhance the clinical efficacy of the used devices. The cohort post market registry represents a novel approach in a way of allowing Clinicians to generate reports based on an evolving controlled and well organized database.

Hypothesis:

Transcatheter Embolization is a recognized primary treatment of various diseases and a viable alternative to existing treatment options. Further that the Registry will foster generation of Consensus Treatment Documents for the benefit of the Clinicians involved in Transcatheter Embolization. Further that the Registry will increase the level of Transcatheter Embolization as a function of Clinicians getting access to data generated in the Registry.

Embolization indications:

The current set-up of the registry focuses on the embolization treatment of visceral arterial aneurysms. In future additional indications for embolization will be added to the scope of the study.

Significance to the scientific field:

A few key opinion leaders in the field of Interventional Radiology (IR), , have identified the need for providing improved clinical evidence on embolization procedures.

There are several factors potentially explain today's limited evidence including:

* rapidly evolving technology,
* absence of consensus on clinical indications/interventional strategy,
* small sample size in term of number of cases/centre/year;
* lack of support from the university/public funding resources as well as the industry,
* low level of required qualification/certification for devices from companies before and during the commercialization process of embolization devices/technologies

All these elements are concurrent toward a need to facilitate independent, high quality, evaluation of clinical outcomes of embolization in a widespread spectrum of applications resulting in publications with a high scientific value and of significance to the healthcare systems.

Registry overview:

A prospective, multi-center, non-randomized cohort registry collecting data of technical and clinical outcome of embolization procedures from participating centers on a standard of care basis.

Duration of the registry:

The estimated duration of the registry is approximately 5 years from the time of first subject enrollment. Subjects will be followed according the standard of care procedures of the participating centers.

Number of sites and subjects:

No limitation has been set on the number of participating sites and subjects. The participating sites will be granted participation approval by one or both co-principal investigators.

Participating investigators:

For physicians and clinical centres to be able to participate in the study they have to be approved by the founders, Marc Sapoval, M.D PhD (Doctor of Philosophy) and Jafar Golzarian, MD and John Kaufman M.D. The founders can name a group of expert as lead principal investigators (LPI) who can represent the founders in each registry.

Only centers and physicians that have the facilities and expertise required for the study can participate in this study.

All participating centers must sign the EmboCoH Charter in order to participate.

EmboCoH is a non for profit organization founded by Marc Sapoval and Jafar Golzarian.

Data Management and Quality Assurance:

The selected platform is e-capture.net. This platform is a property of e-novex. e-novex offers secure and innovative solutions to enhance and conduct e-clinical trials in compliance with the different regulations. e-novex is ISO9001 and ISO27001 certified, ISO is the International Organization for Standardization. The platform is Code of Federal Regulations Title 21, part 11 (21 CFR, part 11) compliant.

Publications and Sharing Data:

Publications will be reviewed by the Steering Committee prior to submission for publication.

EmboCoH will encourage and drive publications in Journals and at Scientific Meetings. EmboCoH will lead the formation of Consensus Documents based on Clinical Outcomes in the database.

Contact information:

Organizational lead:

EmboCoH 17010 40th Place N. Plymouth, MN 55446 (Minnesota) USA EmboCoH is a non for Profit Organization.

Project management:

Gert Andersen gert@transmedicalalliance.com Mob: +45 23 600 650

REGISTRY METHODOLOGY

Registry design:

This is a prospective, multi-center, non-randomized registry. All consecutive subjects eligible for embolization of visceral aneurysms may be included in the registry. Additional indications for embolization may be added to the scope during the course of the registry.

Purpose of the registry:

The purpose of the registry is to provide a worldwide therapeutic embolization data base to provide data and evidence in the field of IR with a focus on embolization and oncology. The data is to be published and can be shared with selected medical and industry professionals.

Primary objective:

The primary objective is collection of initial embolization procedure results and defined as target vessel or lesion occlusion and clinical success.

Secondary objective:

The secondary objective is to collect the organ specific procedural results and outcome.

General inclusion data:

Subjects must meet the following criteria in order to participate within the study:

* Eligible for embolization as defined within the scope of the study.
* Subject (or subject's legally authorized representative) is able and willing to sign the data protection form if and when applicable.

Subject screening & selection:

No specific screening protocol is applicable for the cohort registry. Assessment of patient eligibility is performed as per standard of care and is performed based on data available to the investigator at the time of subject enrollment. Procedure data collection requirements All available data on the initial embolization procedure and organ specific procedure will be collected in the electronic Case Report Form (eCRF).

Follow-up visit data collection:

All subjects will be clinically followed-up as per standard of care of the participating hospital to assess if clinical success was maintained, to evaluate the current health status and whether re-intervention occurred. Imaging follow-up will be included when appropriate and as per standard of care.

It is recommended to have the patients come in for a follow-up visit at one (1), six (6) and 12 months for visceral aneurysms.

Regulatory and Institutional approvals:

The platform is considered to be a non-interventional registry. No formal investigational plan will be created, however available data will be centrally stored outside the hospital and therefore must be compliant with the national or local regulations.

It is the responsibility of each involved center to verify the local requirements prior to the participation. It is strongly recommended to use a written consent form, approved by the relevant institutional review board or ethical committee that confirms the approval of the patient to store anonymous data centrally.

The selected platform is compliant with the overall data protection regulation. Personal access is granted after the approval of the Project Management.

Termination of participation:

All subjects have the right to terminate themselves from participation at any point during the study.

ELIGIBILITY:
Inclusion Criteria:

* Eligible for Embolization and willing to sign Data protection form if required

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with a Visceral Aneurysm
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2014-04; Primary Completion 2019-04 (Estimated); Study Completion 2019-10 (Estimated)

PRIMARY OUTCOMES:
Technical Success (Yes or No) | Assessed within 15 minutes after intervention on the basis of control angiography
  Technical success is defined as occlusion of the target area

SECONDARY OUTCOMES:
Society of Interventional Radiology Classification System for Complications by Outcome - referred to as "SIR Category" (A/B/C/D/E/F) | Assessed within 15 minutes after intervention on the basis of control angiography
  A(No therapy, no consequence)/B (Nominal therapy, no consequence; includes overnight admission for observation only)./C(Require therapy, minor hospitalization (48 hours))/D(Require major therapy, unplanned increase in level of care, prolonged hospitalization)/E(Permanent adverse sequelae)/F(Death)
Occlusion of Aneurysm (Yes or No or Partial) | Assessed within 15 minutes after intervention on the basis of control angiography
  The aneurysm is occlude if no residual blood flow can be observed in the aneurysm.
Immediate Angiographic Complications ('Yes' or 'No' | Assessed within 15 minutes after intervention on the basis of control angiography
  Can be: Migration of the Embolic Material, Vessel dissection or Vessel perforation, Catheter entrapment or Other (that is to be specified)

CONTACTS AND LOCATIONS:
Overall Officials: Jafar Golzarian, MD, Principal Investigator — Unniversity of Minnesota
Locations (1):
- Odense University Hospital, Odense, Denmark